CLINICAL TRIAL: NCT00285805
Title: The Influence of Rosiglitazone on the Diuretic Effect of Furosemide and Amiloride. A Double-blind Placebo Controlled Cross Over Study.
Brief Title: The Influence of Rosiglitazone on the Diuretic Effect of Furosemide and Amiloride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Paul Smits, Radboud University Nijmegen Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AR-49653-3
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2008-10

CONDITIONS: Insulin Resistance
Keywords: Rosiglitazone; Furosemide; Amiloride; Epithelial sodium channel; Sodium excretion
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosiglitazone-placebo (Other)
  Interventions: Drug: Rosiglitazone versus placebo; Drug: response (sodium excretion) to amiloride infusion; Drug: response (sodium excretion) to furosemide infusion
- placebo-rosiglitazone (Other)
  Interventions: Drug: Rosiglitazone versus placebo; Drug: response (sodium excretion) to amiloride infusion; Drug: response (sodium excretion) to furosemide infusion

INTERVENTIONS:
Drug: Rosiglitazone versus placebo
Drug: response (sodium excretion) to amiloride infusion
Drug: response (sodium excretion) to furosemide infusion

SUMMARY:
Thiazolidinedione derivates (TZD's) are Peroxisome-Proliferator-Activated-Receptor-γ agonists (PPARγ-agonists) and enhance insulin sensitivity. One of the side effects, however, is the fact that subjects treated with these drugs seem to be more prone to fluid retention. The precise mechanism of rosiglitazone-related fluid retention is unknown, but it is clear that either primary or secondary renal sodium retention is part of the mechanism. Furthermore in observational studies, TZD-related oedema seems to be resistant to loop diuretic therapy. The recent finding that rosiglitazone induces upregulation of the epithelial sodium channel (ENaC) in the kidney could be the explanation for TZD-related fluid retention and the observed resistance to loop diuretics. In the present human in-vivo study the following hypothesis will be tested:

Rosiglitazone treatment stimulates the activity of ENaC in the distal nephron, which enhances the natriuretic effect of amiloride and decreases the natriuretic effect of furosemide in parallel.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, single-centre, cross-over study with 4 weeks of wash out comparing placebo with rosiglitazone 4 mg bid for 9 weeks treatment periods. Randomization of the treatment sequence will be computer-generated, with a sequentially driven allocation. Randomization and blinding will be performed at the department of Clinical Pharmacy. After 8 (furosemide) and 9 (amiloride) weeks in each period the end-point experiments will be performed. During all visits (week 0, 4, 8, 9) of each period, adverse events and pill compliance will be recorded. In addition, physical examination, foot volume and bio-impedance measurements will be performed and safety chemical, and hematological profiles will be determined. Only at start and at 8 weeks in each period, glucose, insulin and HbA1c are measured. All visits and interventions will be performed at the Clinical Research Center Nijmegen (CRCN).

Furosemide end-point experiment Each participant will attend the hospital at 8 a.m. after an overnight fast and abstinence of alcohol and caffeine for 20 hours, delivering a 24-hour urine collection and the present morning voiding. The previous three days each participant will adhere to an individualized diet containing 150 mmol of sodium and 80 mmol of potassium prescribed by a dietician. First, blood will be collected to measure fasting glucose and insulin concentrations. Then the subject will be given an individualized breakfast including 1 cup of water. Afterwards a brachial vein will be cannulated and connected to a Braunpump (10 ml/hr NaCl 0.9%), followed by blood drawing for safety and vascular hormone measurements (aldosterone, Atrial Natriuretic Peptide (ANP), Brain Natriuretic Peptide (BNP), Vascular Endothelial Growth Factor (VEGF) and renin).

A bolus of furosemide (40 mg) will be injected through a small cannule in a vein of the contra-lateral arm, just after bladder emptying. Venous blood samples will be drawn at 0, 15, 30, 45, 60, 90,120, 150, 180, 240, 300, 360, 420 and 480 minutes after bolus injection to measure plasma furosemide levels. The participants will be asked to urinate regularly, at least hourly. The exact time of voiding and the urine volume will be recorded. Two urine samples will be taken. In one sample, sodium and creatinine concentrations will be measured while the other sample will be light-protected and immediately frozen for measurement of furosemide levels later on. To prevent dehydration each participant will be asked to drink tap water equal to the volume of diuresis in the previous hour. During the test the participant will be sitting on a bed. At noon the participant will be offered an individualized lunch. After 8 hours each participant will leave the hospital with the instruction to adhere to the diet without fluid restrictions and to collect the urine for up to 24 hours after start of the experiment.

Amiloride end-point experiment Until amiloride infusion the procedures will be similar. At time point 0, venous infusion of a loading dose of amiloride will be started (150 μg/kg in 60 minutes) followed by maintenance infusion (0.20 μg/kg/min) for 4 hours. Amiloride will be obtained as a sterile powder in the form of amiloride HCl/2H2O . Directly before use, the powder will be dissolved in NaCl 0,9% up to a concentration of 1 mg/ml and the solution was filtered through a 0.22 μm Millipore filter. Venous blood for measurement of the amiloride concentration will be sampled at 60, 180, 300 and 420 minutes. All the other procedures will be similar to the furosemide experiment.

Pharmacokinetic considerations on the amiloride-dose The peak plasma levels 3-4 hours after intake of 10 or 20 mg amiloride are 20 μg/L (32) and 38-40 μg/L respectively(33). These concentrations are well below the half maximal inhibitory concentration (IC50) of amiloride for Na+/H+ and Na+/Ca2+-transporters and the α1-receptor, but well above the IC50 for ENaC(34). Using the pharmacokinetic characteristics of amiloride(35) we calculated the required amiloride infusion in order to reach a steady-state concentration between 30-45 μg/L.

Exosome extraction:

Urinary exosomes will be isolated by ultracentrifugation and ENaC abundance will be measured by immunoblotting as previously described (19;36) and normalized to urine creatinine levels. 4 µg of protein lysed in Laemmli buffer will be loaded on 8% SDS-PAGE. PAGE, blotting and blocking of the PVDF membranes will be done as previously described. Membrane will be incubated with 1:4000-diluted affinity-purified rabbit α-ENaC antibody (Rossier BC, Lausanne, Switzerland), followed by 1:5,000-diluted goat anti-rabbit IgG's as secondary antibody coupled to horseradish peroxidase. Blotting signals will be visualized using enhanced chemiluminescence. The samples will be normalized for the expression level of α-ENaC in placebo treatment and indicated as percentage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy but with 2 features of the metabolic syndrome (AHA/NHLBI) (16)
* Willing and able to provide a signed and dated written informed consent.
* Male or female subject aged between 30 and 70 years

Exclusion Criteria:

* Fasting glucose > 7,0 mmol/L or the use of hypoglycaemic agents. If fasting plasma glucose is between 6.1 and 7,0 mmol/L,an oral 75 g glucose test will be performed to exclude diabetes mellitus.
* Exposure to a PPAR-g agonist during the last 4 months or a documented significant hypersensitivity to a PPAR-g agonist.
* Participant in another study.
* Angina or heart failure (NYHA I-IV).
* Clinically significant liver disease (3 times the upper normal limit of ALAT, ASAT, AF, γGT or LDH)
* Clinically significant anaemia (male Hb < 6,9 mmol/L, female < 6,25 mmol/L)
* Creatinin clearance < 40 mL/min
* Pregnancy, lactation
* Alcohol or drug abuse. Liquorice

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-02; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Difference in cumulative sodium excretion over an 8-hour period following amiloride infusion after 9 weeks of treatment with either rosiglitazone or placebo. | week: 9, 22

SECONDARY OUTCOMES:
The difference in ER50 (urine excretion rate of furosemide with the half maximal effect) after 8 weeks of treatment with either rosiglitazone or placebo. | week: 8, 21
The difference in the ENac abundance in exosomes in the urine measured after 8 weeks of treatment with either rosiglitazone or placebo | week: 8, 21

CONTACTS AND LOCATIONS:
Overall Officials: Paul Smits, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, head of department Pharmacology and Toxicology.; Cees JJ Tack, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, chairman of the departement of diabetology
Locations (1):
- Radboud University Nijmegen medical centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Nesto RW, Bell D, Bonow RO, Fonseca V, Grundy SM, Horton ES, Le Winter M, Porte D, Semenkovich CF, Smith S, Young LH, Kahn R; American Heart Association; American Diabetes Association. Thiazolidinedione use, fluid retention, and congestive heart failure: a consensus statement from the American Heart Association and American Diabetes Association. October 7, 2003. Circulation. 2003 Dec 9;108(23):2941-8. doi: 10.1161/01.CIR.0000103683.99399.7E. No abstract available. PMID 14662691
- [Background] Hong G, Lockhart A, Davis B, Rahmoune H, Baker S, Ye L, Thompson P, Shou Y, O'Shaughnessy K, Ronco P, Brown J. PPARgamma activation enhances cell surface ENaCalpha via up-regulation of SGK1 in human collecting duct cells. FASEB J. 2003 Oct;17(13):1966-8. doi: 10.1096/fj.03-0181fje. Epub 2003 Aug 15. PMID 12923071
- [Background] Guan Y, Hao C, Cha DR, Rao R, Lu W, Kohan DE, Magnuson MA, Redha R, Zhang Y, Breyer MD. Thiazolidinediones expand body fluid volume through PPARgamma stimulation of ENaC-mediated renal salt absorption. Nat Med. 2005 Aug;11(8):861-6. doi: 10.1038/nm1278. Epub 2005 Jul 10. PMID 16007095
- [Background] Niemeyer NV, Janney LM. Thiazolidinedione-induced edema. Pharmacotherapy. 2002 Jul;22(7):924-9. doi: 10.1592/phco.22.11.924.33626. PMID 12126225
- [Background] van Meyel JJ, Smits P, Russel FG, Gerlag PG, Tan Y, Gribnau FW. Diuretic efficiency of furosemide during continuous administration versus bolus injection in healthy volunteers. Clin Pharmacol Ther. 1992 Apr;51(4):440-4. doi: 10.1038/clpt.1992.44. PMID 1563213
- [Background] Baba WI, Lant AF, Smith AJ, Townshend MM, Wilson GM. Pharmacological effects in animals and normal human subjects of the diuretic amiloride hydrochloride (MK-870). Clin Pharmacol Ther. 1968 May-Jun;9(3):318-27. doi: 10.1002/cpt196893318. No abstract available. PMID 5649984
- [Background] Pisitkun T, Shen RF, Knepper MA. Identification and proteomic profiling of exosomes in human urine. Proc Natl Acad Sci U S A. 2004 Sep 7;101(36):13368-73. doi: 10.1073/pnas.0403453101. Epub 2004 Aug 23. PMID 15326289